CLINICAL TRIAL: NCT00003323
Title: A Phase II Trial of Potency-Sparing Hormonal Therapy in Patients With Elevated Serum PSA After Radiation Therapy or Radical Prostatectomy for Prostate Cancer
Brief Title: Hormone Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9782; U10CA031946 (NIH); CDR0000066274 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-08-13 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer; Sexual Dysfunction and Infertility
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; sexual dysfunction and infertility
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological; Infertility | interventions — Finasteride; Flutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hormone Therapy (Experimental): Treatment of prostate cancer pts post radiation or surgery with potency sparing hormones
  Interventions: Drug: finasteride; Drug: flutamide; Other: quality-of-life assessment

INTERVENTIONS:
Drug: finasteride — 5 mg/d PO
Drug: flutamide — 250 mg PO tid
Other: quality-of-life assessment — Assessment survey administered at baseline, and 3 & 6 months post initiation of treatment

SUMMARY:
RATIONALE: Male hormones can stimulate the growth of prostate cancer cells. Hormone therapy using flutamide and finasteride may fight prostate cancer by reducing the production of male hormones.

PURPOSE: Phase II trial to study the effectiveness of flutamide and finasteride in treating prostate cancer patients with high PSA levels who were previously treated with radiation therapy or radical prostatectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of finasteride and flutamide in suppressing prostate specific antigen (PSA) levels in patients with elevated PSA after definitive radiation therapy or radical prostatectomy for prostate cancer.
* Assess sexual function and other quality of life issues during this therapy.
* Estimate the response to flutamide withdrawal in this group of patients who have not had a major reduction in circulating testosterone levels.
* Measure the response rate to further hormonal manipulation with combined androgen blockade after the failure of this therapy.
* Obtain data that may predict more aggressive disease.

OUTLINE: This is a multicenter study.

Patients receive finasteride and flutamide by mouth three times a day. Patients experiencing recurrence or a greater than 4 nu/mL (above 50%) increase in PSA level will discontinue flutamide treatments. Otherwise, patients continue therapy in the absence of unacceptable toxicity or disease progression.

Quality of life is assessed prior to therapy and at 3 and 6 months.

Patients are followed every 3 months for one year and every 6 months thereafter.

PROJECTED ACCRUAL: This study will accrue 100 patients over 2 years.

ELIGIBILITY:
1. Histologic Documentation: Previous histologic evidence of adenocarcinoma of the prostate.
2. Prior Treatment:

   2.1 Definitive Local Therapy: Patients must have had a previous attempt at definitive therapy, which is defined as a previous radical prostatectomy or radiation therapy with at least 5500 cGy to the prostate.
   1. Patients may have had both radiation therapy to the prostate and surgical resection, given as definitive therapy, provided they began the radiation therapy within 3 months of their prostatectomy. Also, brachytherapy alone and combinations of brachytherapy and external beam radiation therapy are also allowed, if given as a single therapy, and not given for a rising PSA after the previous therapy.
   2. The previous treatment must have occurred at least 6 months, but no more than 10 years, prior to registration.

   2.2 Previous Hormonal Therapy or Other Treatments: Patients may have had no more than 6 months of hormonal therapy with their other treatment, and must have been off all hormones used for the treatment of prostate cancer including Megace for at least 12 months.
   1. No therapy within 2 years with finasteride or other 5 alpha-reductase inhibitors.
   2. No previous chemotherapy for this malignancy.
   3. No orchiectomy.
   4. No corticosteroids in excess of standard replacement doses for adrenal failure.
3. Elevated PSA Criteria:

   3.1 Patients must a PSA level between 1 ng/ml and 10 ng/ml, with a rise of at least 1 ng/ml above the nadir produced by definitive therapy. The PSA level must be repeated at least once, one month later to confirm the rise of 1 ng/ml above nadir.

   3.2 After the second PSA has been drawn to confirm the rise, one additional PSA should be drawn as close to the start of therapy as possible. Therefore, a total of three PSAs must be drawn prior to the start of therapy. Only the last two need to be drawn at the same lab (ie, the second confirmatory PSA and the PSA drawn just prior to the start of the trial). The nadir PSA and the initial PSA suggesting a rise can be drawn at outside laboratories. The combination of the nadir PSA and the two PSAs showing a rise of 1.0 ng/ml are used for determining eligibility. The two elevated PSAs must be at least one month apart.
4. No clear evidence of local recurrence on the digital rectal exam.
5. No metastatic disease on the CT or bone scan.
6. Performance status 0-2
7. Required initial laboratory data

   1. SGOT and/or SGPT ≤2 x upper limits of normal
   2. Creatinine ≤2 x upper limits of normal
   3. Bilirubin ≤2 x upper limits of normal

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 1998-05; Primary Completion 2002-05 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
PSA levels | 1 year post treatment

SECONDARY OUTCOMES:
QOL issues associated with treatment protocol | 3 & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joel Picus, MD, Study Chair — Washington University Siteman Cancer Center
Locations (43):
- United States (43):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Picus J, Halabi S, Small E, et al.: Long term efficacy of peripheral androgen blockade on prostate cancer: CALGB 9782. [Abstract] J Clin Oncol 24 (Suppl 18): A-4573, 2006.
- [Result] Picus J, Halabi S, Small E, et al.: Efficacy of peripheral androgen blockade on prostate cancer: results of CALGB 9782. [Abstract] J Clin Oncol 22 (Suppl 14): A-4559, 396s, 2004.
- [Result] Picus J, Halabi S, Hussain A, et al.: Efficacy of peripheral androgen blockade on prostate cancer: initial results of CALGB 9782. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-727, 2002.